CLINICAL TRIAL: NCT06878053
Title: Benefit of Ethanol Sclerotherapy of Endometriomas Before Ovarian Stimulation on Pregnancy Rates in IVF/ICSI
Acronym: SCLERENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Nelly SWIERKOWSKI-BLANCHARD, MD, MD, Poissy-Saint Germain Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A02459-38
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Infertile Women Undergoing IVF or ICSI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ethanol sclerotherapy group (Experimental)
  Interventions: Procedure: ethanol sclerotherapy
- group without intervention (No Intervention)

INTERVENTIONS:
Procedure: ethanol sclerotherapy — The originality of this project consists in evaluating the effectiveness of ethanol sclerotherapy of endometrioma(s) in infertile patients before IVF/ICSI, excluding patients who have previously had an ovarian cystectomy. To date, no prospective randomized comparative study between ethanol sclerotherapy of endometriomas and therapeutic abstention has been carried out.
  Arms: ethanol sclerotherapy group

SUMMARY:
Evaluation of progressive pregnancy rates (with an embryo with cardiac activity at 12 weeks), on a first attempt at IVF/ICSI (fresh and frozen embryo transfers) following the discovery of one or two endometrioma(s) of 30 to 80 mm, without a history of cystectomy, and comparison between the two groups: ethanol sclerotherapy and therapeutic abstention

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged 18 to 43,
* Presenting one or 2 endometriotic cysts of 30 mm to 80 mm long axis, confirmed by ultrasound and/or pelvic MRI and without signs of atypia,
* With indication of IVF/ICSI, first IVF/ICSI after the discovery of endometriosis cyst(s),
* Having given their consent.

Exclusion Criteria:

* A history of ovarian cystectomy,
* A non-homogeneous cyst that cannot be punctured (risk of incomplete aspiration),
* Complex adnexal image that cannot exclude an associated hematosalpinx (communicating hematosalpinx, tissue component),
* A recent tubo-ovarian infection,
* An active, untreated vaginal infection,
* Anticoagulant treatment at a therapeutic dose,
* All adult patients protected by law (under guardianship or curatorship),
* Problems understanding the French language,
* Participation in intervention research,
* All patients not affiliated to the social security system.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 174 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
cumulative rate of active pregnancies | 12 weeks
  Cumulative rate of active pregnancies defined by the presence of an embryo with cardiac activity at 12 weeks per IVF/ICSI cycle, including fresh and frozen embryo transfers in an IVF/ICSI attempt.

IPD SHARING:
Plan to Share IPD: Undecided